CLINICAL TRIAL: NCT01929720
Title: Worry, Uncertainty and Insomnia: A Cognitive-behavioral Intervention for Cancer Survivors
Brief Title: Cognitive-Behavioral Intervention for Worry, Uncertainty, and Insomnia for Cancer Survivors
Acronym: FOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other); Lance Armstrong Foundation (Other)
Responsible Party: Principal Investigator, Sharla Wells-Di Gregorio, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-09096; NCI-2012-02879 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-13; First posted 2013-08-28 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Anxiety Disorder; Worry; Uncertainty; Sleep Disorders; Insomnia; Fatigue; Pain; Depression; Cognitive-behavioral Therapy; Psychological Intervention; Esophageal Cancer; Pancreatic Cancer; Leukemia; Lung Cancer; Multiple Myeloma; Ovarian Neoplasm; Stage III or IV Cervical or Uterine Cancer; Stage IIIB, IIIC, or IV Breast Cancer; Glioblastoma Multiforme; Relapsed Lymphoma; Stage III or IV Colorectal Cancer; Stage IIIC or IV Melanoma
Keywords: cancer; cancer survivors; worry; insomnia; symptoms; fatigue; depression; anxiety
MeSH Terms: conditions — Anxiety Disorders; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Fatigue; Pain; Depression; Esophageal Neoplasms; Pancreatic Neoplasms; Leukemia; Lung Neoplasms; Multiple Myeloma; Ovarian Neoplasms; Uterine Neoplasms; Glioblastoma; Lymphoma; Neoplasms | interventions — Cognitive Behavioral Therapy; Uncertainty; Acceptance and Commitment Therapy; Psychosocial Intervention; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (CBT for worry, uncertainty & insomnia) (Experimental): Patients wear a wrist actigraph and complete a sleep diary and worry record daily in weeks 1 and 5. Patients participate in a Behavioral Intervention (cognitive-behavioral therapy) in which they receive education on the components of anxiety (physical cognitive, and behavioral) and practice relaxation techniques and behavioral sleep strategies in weeks 2-5.
  Interventions: Behavioral: Cognitive-behavioral therapy for worry, uncertainty & insomnia
- Arm II (wait-list control) (Active Comparator): Patients wear a wrist actigraph and complete a sleep diary and worry record daily in weeks 1 and 5. This is a wait-list comparison, so after six weeks, patients in the control group complete the behavioral (cognitive-behavioral therapy)intervention for worry, uncertainty, and insomnia.
  Interventions: Behavioral: Cognitive-behavioral therapy for worry, uncertainty & insomnia

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy for worry, uncertainty & insomnia — This intervention involves teaching the participant in-person strategies for managing worry, uncertainty, and insomnia and involves home practice.
  Other Names: Cognitive-behavioral Therapy; Acceptance and Commitment Therapy; Psychological Intervention; Behavior Therapy; Behavioral Modification; Behavioral Therapy; Behavioral Treatment

SUMMARY:
This randomized clinical trial studies a cognitive-behavioral intervention to treat worry, uncertainty, and insomnia in cancer survivors. Counseling may reduce anxiety and insomnia as well as improve the well-being and quality of life of cancer survivors. This study also explores the neuro-immunologic correlates of anxiety and insomnia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To complete a randomized pilot trial of a cognitive-behavioral anxiety-insomnia intervention to determine the impact of this intervention on patient worry, intolerance of uncertainty, and sleep efficiency.

II. Explore the underlying endocrine and immune mechanisms responsible for a specific symptom cluster (anxiety-insomnia-depression-pain-fatigue) observed among advanced cancer patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients wear a wrist actigraph, collect saliva samples, and complete a sleep diary and worry record daily in weeks 1 and 5. Patients also receive education on the components of anxiety (physical cognitive, and behavioral) and practice relaxation techniques and behavioral sleep strategies in weeks 2-5. Blood draw is optional.

ARM II: Patients wear a wrist actigraph, collect saliva samples, and complete a sleep diary and worry record daily in weeks 1 and 5. Blood draw is also optional. This is a wait-list control arm, so patients in this arm, after a six-week period of treatment as usual with their oncologist, then receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* stage III or IV colorectal cancer
* pancreatic cancer
* esophageal cancer
* multiple myeloma
* leukemia
* stage IIIC and IV melanoma
* ovarian cancer
* stage III & IV cervical cancer
* stage III & IV uterine cancer
* stage IIIB, IIIC, and IV breast cancer
* glioblastoma multiforme
* early relapse (< 1 year) lymphoma

Exclusion Criteria:

* co-morbid immunologic disease (i.e. rheumatoid arthritis, systemic lupus)
* neurologic disease (i.e. multiple sclerosis, Parkinson's, Alzheimer's) that would affect neuro-immune assessment or completion of study questionnaires
* mania (if patient has bipolar disorder)
* active substance abuse disorders such as alcohol dependence and cocaine abuse will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in worry on the Penn State Worry Questionnaire | From baseline to 6 weeks
  A linear mixed model will be used to evaluate the change from pre to post on the Penn State Worry Questionnaire. The model will include group (treatment vs. control), time (pre vs. post), and group-time interaction effects. If the outcome measure is not normally distributed with equal variance across groups, then the outcomes will be log transformed in order to meet these assumptions for the mixed models.
Changes in sleep efficiency on the Insomnia Severity Index | From baseline to 6 weeks
  A linear mixed model will be used to evaluate the change from pre to post on the Insomnia Severity Index. The model will include group (treatment vs. control), time (pre vs. post), and group-time interaction effects. If the outcome measure is not normally distributed with equal variance across groups, then this outcome will be log transformed in order to meet these assumptions for the mixed models.
Changes in intolerance of uncertainty on the Intolerance of Uncertainty Scale | From baseline to 6 weeks
  A linear mixed model will be used to evaluate the change from pre to post on the Intolerance of Uncertainty Scale . The model will include group (treatment vs. control), time (pre vs. post), and group-time interaction effects. If the outcome measure is not normally distributed with equal variance across groups, then the outcome will be log transformed in order to meet these assumptions for the mixed models.

SECONDARY OUTCOMES:
Levels of cortisol | Baseline
  This is an exploratory hypothesis. We are using only baseline data to estimate the correlation between the continuous anxiety scale (STAI scores range from 20 - 80) and plasma and serum cortisol.
Levels of pro and anti-inflammatory cytokines | Baseline
  This is an exploratory hypothesis. We are using only baseline data to estimate the correlation between the continuous anxiety scale (STAI scores range from 20 - 80) and pro and anti inflammatory cytokines.
Levels of myeloid-derived suppressor cells (MDSC) | Baseline
  This is an exploratory hypothesis. We are using only baseline data to estimate the correlation between the continuous anxiety scale (STAI scores range from 20 - 80) and myeloid-derived suppressor values.

CONTACTS AND LOCATIONS:
Overall Officials: Sharla Wells-Di Gregorio, Ph.D., Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Wexner Medical Center at The Ohio State University Department of Psychiatry, Columbus, Ohio, United States

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Wells-Di Gregorio S, Flowers S, Peng J, Marks DR, Probst D, Zaleta A, Benson D, Cohn DE, Lustberg M, Carson W, Magalang U, Baltimore S, Ancoli-Israel S. Combined Treatment With Cognitive Behavioral Therapy for Insomnia and Acceptance and Commitment Therapy Enhances Objective and Subjective Reports of Sleep in Patients With Advanced Cancer. Psychooncology. 2025 Apr;34(4):e70141. doi: 10.1002/pon.70141. PMID 40204663
- See also: Center for Palliative Care — http://palliativecare.osu.edu/research/